CLINICAL TRIAL: NCT07204145
Title: The Efficacy of Laser Acupuncture for Behavioral and Psychological Symptoms of Dementia: A Randomized Controlled Trial
Brief Title: Laser Acupuncture for Behavioral and Psychological Symptoms of Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH114-REC3-115
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Behavioral and Psychological Symptoms of Dementia (BPSD); Dementia
Keywords: Dementia; Behavioral and Psychological Symptoms of Dementia (BPSD); Laser Acupuncture
MeSH Terms: conditions — Behavior; Dementia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a parallel design to one of three groups: laser acupuncture, sham laser acupuncture, or usual care. The interventions will be delivered concurrently, and outcomes will be assessed at baseline and five follow-up time points.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers, and outcome assessors will be masked to group assignment. The investigator delivering the intervention will be aware of the assignment due to the nature of the laser acupuncture procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Acupuncture (Experimental): Participants receive laser acupuncture with an 808 nm laser pen at GV20, ST36, and PC6, three times per week, 10 seconds per acupoint.
  Interventions: Device: Laser Acupuncture (808 nm laser pen)
- Sham Laser Acupuncture (Placebo Comparator): Participants receive sham laser acupuncture with the same procedure but without active laser output.
  Interventions: Device: Sham Laser Acupuncture
- Usual Care (No Intervention): Participants receive standard dementia care provided by the facility, including routine medical treatment, nursing care, and daily support, without additional acupuncture or laser intervention.

INTERVENTIONS:
Device: Laser Acupuncture (808 nm laser pen) — Participants receive laser acupuncture using an 808 nm, 100 mW semiconductor laser pen applied at acupoints GV20, bilateral ST36, and bilateral PC6. Each acupoint is irradiated for 10 seconds, three times per week, for 12 weeks.
  Arms: Laser Acupuncture
Device: Sham Laser Acupuncture — Participants receive the same procedure as the laser acupuncture group, using an 808 nm semiconductor laser pen applied at acupoints GV20, bilateral ST36, and bilateral PC6. The device is identical in appearance and produces lights and beeping sounds; however, it delivers no energy output. Each acupoint is contacted for 10 seconds, three times per week, for 12 weeks.
  Arms: Sham Laser Acupuncture

SUMMARY:
This study uses a laser acupuncture pen to stimulate specific acupoints, aiming to evaluate its effectiveness in improving behavioral and psychological symptoms of dementia (BPSD).

DETAILED DESCRIPTION:
Participants will be dementia patients residing in institutions who present with BPSD symptoms. A laser acupuncture pen with a wavelength of 808 nm will be used to irradiate the following acupoints three times per week: GV20, ST36, and PC6, with each acupoint irradiated for 10 seconds per session. The severity of BPSD, activities of daily living, and cognitive function will be assessed using the NPI, MMSE, and ADL scales, respectively, while recording the dosage of oral Psychotropic medicationsmedications. A total of six assessments, including the baseline, will be conducted to evaluate the immediate, short-term, and long-term effects of laser acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Dementia: Participants must have a clinical diagnosis of dementia, of any type or severity
* Consent: Written informed consent provided by the participant's family or legal representative.

Exclusion Criteria:

* Refusal to sign the informed consent form.
* Unable to cooperate with the intervention procedure despite repeated attempts.
* History of epilepsy.
* End-stage liver disease.
* End-stage renal disease requiring hemodialysis.
* Presence of brain tumor or history of major brain surgery.
* Acute cardiovascular or cerebrovascular events within the past 3 months (e.g., unstable angina, myocardial infarction, stroke).
* Use of a cardiac pacemaker.
* Currently receiving acupuncture or traditional Chinese medicine treatment.
* Presence of acute illness.
* Abnormal blood pressure or fever.
* Presence of malignant tumor.
* Pregnancy.
* Presence of unusual physical abnormalities or sensory nerve disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) total score | Baseline (before intervention), 1 week after first intervention, 1 month after first intervention, 2 months after first intervention, 3 months after first intervention, and 4 months after first intervention (also 1 month after the end of intervention)
  The Neuropsychiatric Inventory (NPI) assesses behavioral and psychological symptoms of dementia. The NPI total score ranges from 0 to 144, with higher scores indicating more severe symptoms (worse outcome).

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) total score | Baseline (before intervention), 1 week after first intervention, 1 month after first intervention, 2 months after first intervention, 3 months after first intervention, and 4 months after first intervention ( also 1 month after the end of intervention).
  The Mini-Mental State Examination (MMSE) assesses global cognitive function. The MMSE total score ranges from 0 to 30, with higher scores indicating better cognitive performance (better outcome).
Activities of Daily Living (ADL) total score | Baseline (before intervention), 1 week after first intervention, 1 month after first intervention, 2 months after first intervention, 3 months after first intervention, and 4 months after first intervention ( also 1 month after the end of intervention).
  The Activities of Daily Living (ADL) scale evaluates functional independence in daily activities such as feeding, bathing, dressing, mobility, and continence. Scoring is based on the Barthel Index method, with a total score ranging from 0 to 100. Higher scores indicate greater independence in daily activities (better outcome).
Change in psychotropic medication use | Baseline (before intervention), 1 week after first intervention, 1 month after first intervention, 2 months after first intervention, 3 months after first intervention, and 4 months after first intervention (also 1 month after the end of intervention).
  Tracks changes in the dosage and number of prescribed psychotropic medications, including antipsychotics, antidepressants, anxiolytics, and hypnotics.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchen Lee, MD, PhD, Principal Investigator — Principal Investigator, Department of Acupuncture
Locations (2):
- Taiwan (2):
  - Taoyuan Veteran's Home, Taoyuan, Bade District
  - China Medical University Hospital, Taichung, Taichung City

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been determined. Any decision regarding data sharing will require careful consideration of participant privacy and data protection, particularly for individuals with dementia.